CLINICAL TRIAL: NCT03293277
Title: A Phase I Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Intranasal Dexmedetomidine in Healthy Subjects
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of Intranasal Dexmedetomidine in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR0171401-101
Record Dates: First submitted 2017-08-23; First posted 2017-09-26 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Sedation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A1 (Experimental): 20µg Dexmedetomidine or Placebo is administered intranasally on Day 1, and 20µg Dexmedetomidine or Placebo is administered intravenousally on Day 8
  Interventions: Drug: Intranasal Dexmedetomidine; Drug: Intravenous Dexmedetomidine; Drug: Intranasal Placebo; Drug: Intravenous Placebo
- A2 (Experimental): 20µg Dexmedetomidine or Placebo is administered intravenousally on Day 1, and 20µg Dexmedetomidine or Placebo is administered intranasally on Day 8
  Interventions: Drug: Intranasal Dexmedetomidine; Drug: Intravenous Dexmedetomidine; Drug: Intranasal Placebo; Drug: Intravenous Placebo
- B1 (Experimental): 40µg Dexmedetomidine or Placebo is administered intranasally on Day 1, and 40µg Dexmedetomidine or Placebo is administered intravenousally on Day 8
  Interventions: Drug: Intranasal Dexmedetomidine; Drug: Intravenous Dexmedetomidine; Drug: Intranasal Placebo; Drug: Intravenous Placebo
- B2 (Experimental): 40µg Dexmedetomidine or Placebo is administered intravenousally on Day 1, and 40µg Dexmedetomidine or Placebo is administered intranasally on Day 8
  Interventions: Drug: Intranasal Dexmedetomidine; Drug: Intravenous Dexmedetomidine; Drug: Intranasal Placebo; Drug: Intravenous Placebo
- C (Experimental): 80µg Dexmedetomidine or Placebo is administered intranasally on Day 1
  Interventions: Drug: Intranasal Dexmedetomidine; Drug: Intranasal Placebo

INTERVENTIONS:
Drug: Intranasal Dexmedetomidine — Intranasal Dexmedetomidine
Drug: Intravenous Dexmedetomidine — Intravenous Dexmedetomidine
  Arms: A1; A2; B1; B2
Drug: Intranasal Placebo — Intranasal Placebo
Drug: Intravenous Placebo — Intravenous Placebo
  Arms: A1; A2; B1; B2

SUMMARY:
The aim of this study is to investigate the safety, pharmacokinetics, pharmacodynamics of intranasal dexmedetomidine, and comparative pharmacokinetics of intranasally and intravenously administered dexmedetomidine in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male 18 - 40 years of age
* Body weight >/= 50 kg (male) or >/= 45 kg (female), with BMI between 19.0 and 26.0 kg/m2, inclusive
* Capable of giving written informed consent

Exclusion Criteria:

* Clinically significant disease or conditions that may place the subject at unacceptable risk as a participant in the study, or that may interfere with the safety, tolerability or pharmacodynamic evaluations in the study
* Laboratory tests positive for HIV, Hepatitis B virus surface antigen, or Hepatitis C virus antibody; positive drug or alcohol test
* Major surgery within 4 weeks of screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Baseline to 7 days after dose administration
  Number of subjects with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China